CLINICAL TRIAL: NCT02455856
Title: A Study to Investigate the Potential Effects of Repeated Administration of Itraconazole on the Pharmacokinetics of JNJ-42847922 in Healthy Male Subjects
Brief Title: Study to Investigate Effects of Repeated Administration of Itraconazole on Pharmacokinetics of JNJ-42847922 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Cilag N.V./S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR107144; 42847922EDI1005 (Other: Janssen Cilag N.V./S.A., Belgium); 2014-005499-27 (EudraCT Number)
Record Dates: First submitted 2015-05-26; First posted 2015-05-28 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Healthy
Keywords: Healthy; Itraconazole; JNJ-42847922
MeSH Terms: interventions — seltorexant; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (1):
- JNJ-42847922 plus Itraconazole (Experimental): Participants will receive single dose of 5 milligram (mg) JNJ-42847922 as 5 mg/milliliter [mL] oral solution on Day 1 and Day 6 and itraconazole as 200 mg (2*100 mg capsule) from Day 2 to Day 6.
  Interventions: Drug: JNJ-42847922; Drug: Itraconazole

INTERVENTIONS:
Drug: JNJ-42847922 — Participants will receive single dose of 5 milligram (mg) JNJ-42847922 as 5 mg/milliliter [mL] oral solution on Day 1 and Day 6.
Drug: Itraconazole — Participants will receive single dose of itraconazole as 200 mg (2*100 mg capsule) from Day 2 to Day 6.

SUMMARY:
The purpose of this study is to assess the effects of repeated once daily administration of 200 milligram (mg) of itraconazole (steady state) on the single-dose pharmacokinetics of JNJ 42847922 in healthy, male participants.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), fixed-sequence, single-center, single-dose study designed to assess the effects of steady-state itraconazole exposure on the pharmacokinetics of a single oral dose of JNJ 42847922 in healthy male participants. The duration of study will be approximately of 6 weeks per participant. The study consists of 3 parts: Screening (that is, 21 days before study commences on Day 1); Open-label Treatment (6 days); and Follow-up (7 to 14 days after last dose of study drug or early withdrawal).

All eligible participants will receive single oral doses of 5 milligram (mg) JNJ-42847922 on Day 1 and Day 6. A daily dose of 200 mg itraconazole will be administered from Day 2 to Day 6. Followed by an overnight fast of at least 8 hours participants will be administered with study treatment 30 minutes after light breakfast. Participants will not be allowed to have food until 4 hours of drug administration. Blood samples will be collected for evaluation of pharmacokinetics at pre-dose and post-dose of study treatment. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants aged between 18 and 55 years, inclusive
* Body mass index (BMI) between 18 and 30 kilogram/meter^2 inclusive (BMI = weight/height^2)
* Nonsmoker (not smoked for at least 3 months prior to screening)
* Men who are sexually active with a woman of childbearing potential and have not had a vasectomy must agree to use a barrier method of birth control e.g., either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study and for 3 months after receiving the last dose of study drug. In addition, their female partners should also use an appropriate method of birth control for at least the same duration
* Participants must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study and comply with the study procedures and restrictions

Exclusion Criteria:

* Clinically significant abnormal values for hematology, clinical chemistry or urinalysis at screening or admission
* Clinically significant abnormal physical examination, vital signs or 12-lead ECG at screening, on Day -1 or on Day 1, predose
* History of or current significant psychiatric and other illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematological disease, lipid abnormalities, bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, Parkinson's disease, infection, or any other illness that the Investigator considers should exclude the subject. History of epilepsy or fits or unexplained black-outs
* Serology positive for hepatitis B surface antigen (HBsAg), hepatitis C antibodies (HCV) or human immunodeficiency virus (HIV) antibodies
* History of clinically significant drug and/or food allergies

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-05-18 (Actual); Primary Completion 2015-06-19 (Actual); Study Completion 2015-06-19 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of JNJ-42847922 | up to Day 6
  The Cmax is the maximum plasma concentration.
Time to Reach Maximum Concentration (tmax) of JNJ-42847922 | up to Day 6
  The tmax is time to reach the maximum observed plasma concentration.
Time to Reach Last Quantifiable Plasma Concentration (tlast) of JNJ-42847922 | up to Day 6
  The tmax is time to last observed quantifiable plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) of JNJ-42847922 | up to Day 6
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of JNJ-42847922 | up to Day 6
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z), wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time; C(last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Area Under the Plasma Concentration-Time Curve From Time Zero to 24 Hours (AUC [0-24]) of JNJ-42847922 | up to Day 6
  The AUC (0-24) is the area under the plasma concentration-time curve from time 0 to time 24 hours
Elimination Half-Life (t [1/2] Lambda) of JNJ-42847922 | up to Day 6
  Elimination half-life (t [1/2] Lambda) is associated with the terminal slope (lambda [z]) of the semi logarithmic drug concentration-time curve, calculated as 0.693/lambda(z).
Rate Constant (Lambda[z]) | up to Day 6
  Lambda(z) is first-order rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Apparent total body clearance (CL/F) of JNJ-42847922 | up to Day 6
  Clearance is a quantitative measure of the rate at which a drug substance is removed from the body. The CL/F will be calculated by dividing the dose by AUC (0-infinity)
Apparent volume of distribution at the terminal Phase (Vd[z] /F) of JNJ-42847922 | up to Day 6
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug.The Vd(z)/F will be calculated by dividing CL/F by lambda(z).
Mean Residence Time of JNJ-42847922 | up to Day 6
  Mean residence time, calculated as area under the first moment curve (AUMC[0-infinity]/AUC(0-infinity).
Amount of JNJ-42847922 Excreted in Urine (Ae) | up to Day 6
  amount excreted into the urine, calculated by multiplying the urinary volume with the urinary concentration.
Percentage of JNJ-42847922 Dose Excreted in Urine | up to Day 6
  Amount excreted into the urine, expressed as a percentage of the administered dose, calculated as [Ae/dose]*100, and corrected for molecular weight when necessary.
Renal Clearance | up to Day 6
  Renal clearance calculated as Ae (total)/AUC (infinity).

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | up to End of study (7 to 14 days after lasr dose of study drug or early withdrawal)
  An AE was any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Locations (1):
- Berlin, Germany